CLINICAL TRIAL: NCT01186653
Title: Effect of High Dose Inhaled Budesonide and Fluticasone on Adrenal Function in Patients With Moderate to Severe COPD
Brief Title: Effect on Adrenal Function of Budesonide Versus Fluticasone in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: James Illingworth, Hull and East Yorkshire Hospitals Trust
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AcadMedCTU030406
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide, Formoterol Fumarate Drug Combination; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Symbicort (Experimental): Symbicort® (budesonide / formoterol, 400 micrograms/9 micrograms one puff bd, dose as per NICE guidelines
  Interventions: Drug: budesonide / formoterol
- Seretide (Active Comparator): fluticasone/salmeterol, 250 micrograms/25 micrograms two puffs bd, dose as per NICE guidelines
  Interventions: Drug: fluticasone/salmeterol

INTERVENTIONS:
Drug: budesonide / formoterol — budesonide / formoterol, 400 micrograms/9 micrograms one IH bd
  Other Names: Symbicort
  Arms: Symbicort
Drug: fluticasone/salmeterol — fluticasone/salmeterol, 250 micrograms/25 micrograms two puffs bd, dose as per NICE guidelines
  Other Names: Seretide
  Arms: Seretide

SUMMARY:
National Institute for Clinical Excellence (NICE) guidelines recommend high dose inhaled steroids for patients with moderate to severe Chronic Obstructive Pulmonary Disease (COPD, a common chronic disease related to smoking) who are having two or more exacerbations requiring treatment with antibiotics or oral steroids in a 12 month period. The preparations licensed for this indication commercially available are Symbicort® and Seretide®. High dose inhaled steroids (contained in both) can cause suppression of the adrenal glands. The investigators want to assess adrenal suppression caused by the two preparations and compare. The results could guide investigators in prescribing these preparations.

DETAILED DESCRIPTION:
Background COPD is a very common disease which is chronic and progressive. Current NICE guidelines recommend the use of inhaled steroid in relatively high dose in patients with moderate to severe disease who are having two or more exacerbations requiring treatment with antibiotics or oral steroids in a 12 month period.The aim of this treatment is to reduce the exacerbation rates and slow decline in health status. None of the inhaled steroids currently available are licensed for use alone in the treatment of COPD. They are prescribed in combination with a long acting beta 2 agonist (LABA, a medication which leads to dilatation of the airways), which is an effective combination. The combination of a LABA with inhaled steroid preparations available includes Symbicort® (containing budesonide and formoterol fumarate and Seretide® (containing fluticasone propionate and salmeterol xinafoate). Symbicort® has been evaluated in randomized controlled in patients with COPD and has been found to be beneficial compared to either component alone. Similar data is available for Seretide® as well. There are no large trials directly comparing the two different preparations and quite often the choice between the two is made rather empirically. Although inhaled steroids have a very good safety profile at low doses, the dose used in both these preparations for use in COPD is high and has got potential for adverse effects such as adrenal (a gland in the body which secretes steroids) suppression. Studies have shown that marked adrenal suppression occurs with high dose inhaled steroids.However the doses used in various studies have been different and these studies have been in the asthmatic group of patients, the response of whom may be different from those with COPD. The effect of adrenal function can be assessed by a simple analysis of an overnight urine sample collection. It is difficult to decide which of the treatments to choose on initiation of therapy. We wish to compare the adrenal suppression between the two treatments and determine whether there is any difference, which could influence decision on treatment in specific patient groups who are considered more at risk for adverse effects. Study design This study will be conducted at a single centre. The investigators will be responsible for the study. The study is designed as an 8 week study in which patients will cross over from one arm of the study group to another. Patients with COPD who are on current treatment with either Symbicort® or Seretide® on doses as per NICE guidelines will be included. The treatment doses are Symbicort® (budesonide / formoterol, 400 micrograms/9 micrograms) one puff bd and Seretide® (fluticasone/salmeterol, 250 micrograms/25 micrograms) two puffs bd. We plan to include 30 patients either on current treatment with Symbicort® or Seretide®. On visit 1 : Patients would either be on treatment with high dose Symbicort® OR Seretide® (on treatment for at-least four weeks). The patients will be re-trained in the correct use of their current inhaler and re-educated has to how often they should be taking the medication. The patient will be guided to take the treatment as indicated for 4weeks, at the end of the 4 week treatment they will be asked to collect an overnight (12 hrs) urine sample (21:00 hrs-09:00hrs). The patient will return to the clinic for visit 2 where they will return the urine sample and quality of life in the previous 4 weeks will be assessed by means of a modified St Georges Respiratory questionnaire. If the patient was on treatment with Symbicort® it will be switched over to Seretide® and vice-versa. The patient will be seen 4 weeks later on visit 3.

A bottle for collecting an overnight ( 12 hours) urine sample will be given to the patient for urine collection at the end of the 4 week treatment period. On visit 3: the patient will return the overnight urine sample and The quality of life of the patient in the previous 4 weeks will be assessed using the modified St Georges Respiratory Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of COPD.
* Criteria for treatment with inhaled steroids met as per NICE guidelines.
* Patients on treatment with either Symbicort® or Seretide® at the time of recruitment (on treatment dose as per NICE guidelines).
* Recruited patients are able to understand and co-operate with the study conduct and are willing to give written consent.

Exclusion Criteria:

* Patients with any concomitant disease which may interfere with the study procedure or evaluation.(self explanatory)
* A recent exacerbation of COPD within the last 8 weeks.( will interfere with assessment )
* Use of oral steroids within the last 2 months.(will interfere with assessment)
* Use of ocular, intra-articular, rectal or other steroids during 4 weeks prior to inclusion.(will interfere with assessment)
* Participation in any other study (use of investigational product) within 4 weeks prior to inclusion.(potential to interfere with assessment)
* Alcohol or drug abuse.(will interfere with assessment)
* Inability to follow study procedures.(self explanatory)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Overnight urinary cortisol:creatinine ratio | 12 hr
  The primary objective of the study is to determine any change in overnight urinary cortisol:creatinine ratio from that measured after 4 weeks treatment with high dose Symbicort® (budesonide / formoterol, 400 micrograms/9 micrograms one puff bd, dose as per NICE guidelines) to that following 4 weeks treatment with Seretide® (fluticasone/salmeterol, 250 micrograms/25 micrograms two puffs bd, dose as per NICE guidelines)

SECONDARY OUTCOMES:
Quality of life | 4 week
  Secondary objective is to compare quality of life as measured with a modified St Georges respiratory Questionnaire with high dose Symbicort® (budesonide / formoterol, 400 micrograms/9 micrograms one puff bd, dose as per NICE guidelines) and Seretide® (fluticasone/salmeterol, 250 micrograms/25 micrograms two puffs bd, dose as per NICE guidelines)

CONTACTS AND LOCATIONS:
Overall Officials: Alyn H Morice, Professor, Principal Investigator — Hull and East Yorkshire NHS Trust
Locations (1):
- Respiratory Medicine, Castgle Hill Hospital, Cottingham, East Yorkshire, United Kingdom